CLINICAL TRIAL: NCT01818869
Title: A Phase 1, Single Centre, Double-blind, Randomised, Placebo-controlled, Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics After Administration of Multiple Ascending (MAD) Once Weekly Inhaled Doses of AZD8848 in Healthy Subjects
Brief Title: To Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Doses AZD8848 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: D0542C00002
Record Dates: First submitted 2013-03-18; First posted 2013-03-27 (Estimated); Last update posted 2015-08-14 (Estimated); Status verified 2015-08

CONDITIONS: Safety,; Tolerability,; Healthy Subjects
Keywords: Safety,; tolerability,; Phase I,; pharmacokinetic,; pharmacodynamic,; inhaled
MeSH Terms: conditions — Respiratory Aspiration | interventions — AZD8848

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AZD8848 (Experimental): Subjects will participate in 1 of 3 groups and receive multiple doses of AZD8848 or matching placebo In each group 6 subjects will receive AZD8848 and 2 subjects will receive matching placebo.
  Interventions: Drug: AZD8848
- Placebo to match AZD8848 (Placebo Comparator): Subjects will participate in 1 of 3 groups and receive multiple doses of AZD8848 or matching placebo. In each group 6 subjects will receive AZD8848 and 2 subjects will receive matching placebo.
  Interventions: Drug: Placebo to match AZD8848

INTERVENTIONS:
Drug: AZD8848 — Multiple doses inhaled IMP via a nebulizer
  Arms: AZD8848
Drug: Placebo to match AZD8848 — Multiple doses inhaled matching placebo via a nebulizer
  Arms: Placebo to match AZD8848

SUMMARY:
This study will investigate the safety, tolerability, pharmacokinetics and pharmacodynamics of multiple ascending doses of AZD8848 in healthy subjects.

DETAILED DESCRIPTION:
A Phase 1, Single Centre, Double-blind, Randomised, Placebo-controlled, Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics after Administration of Multiple Ascending (MAD) Once Weekly Inhaled Doses of AZD8848 in Healthy Subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects aged 18 to 50 years (inclusive) with suitable veins for cannulation or repeated venipuncture
* Women must be of non-childbearing potential or must have been stable on a highly effective contraceptive for at least 3 months prior to Screening and be willing to continue on the chosen contraceptive with additonal use of condom until 3 months postdose
* Male subjects should be willing to use barrier contraception ie, condoms, from the first day of investigational product administration until 3 months after the last administration of investigational product
* Have a body mass index (BMI) between 18 and 32 kg/m2 and weigh at least 50 kg and no more than 110 kg
* Women must have a negative pregnancy test at screening and on admission to the study centre, must have a date of last menstruation, must not be lactating or must be of non-childbearing potential

Exclusion Criteria:

* Abnormal vital signs, after 10 minutes supine rest, defined as any of the following: SBP >140 mmHg, Diastolic blood pressure (DBP) >90 mmHg, Heart rate <40 or >85 beats per minute
* History of asthma or allergic rhinitis
* Prolonged QTcF >450 ms or shortened QTcF <340 ms or family history of long QT syndrome
* History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the Investigator or history of hypersensitivity to drugs with a similar chemical structure or class as AZD8848 - Any clinically significant abnormalities in clinical chemistry.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2014-01; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline up to 77 days in safety variables (adverse events, vital signs, body temperature, physical exams, ECGs, clinical laboratory tests, pulse oximetry, spirometry). | From screening visit (Day -42) through the Treatment Follow Up visit (Day 35) at multiple timepoints up to 77 days.

SECONDARY OUTCOMES:
Single dose pharmacokinetics profile for AZD8848 and its acid metabolite (AZ12432045) combined and, if possible, for AZD8848 alone in plasma and urine from healthy subjects | Plasma: From Days 1 and 22, pre-dose, 5, 10, 20, 30, 45, 60, 90 min, 2, 3, 4, 6, 8 and 24 hrs post dose. Urine: From days 1 and 22, pre-dose, 0 to 6, 6 to 12 and 12 to 24 hrs post dose
  PK parameters: Cmax, tmax, area under the plasma concentration-time curve from zero to 24 hours postdose (AUC(0-24)), from zero to the time of the last quantifiable concentration (AUC(0-t)) and from zero to infinity (AUC), CL/F, Vz/F, CLR and Ae
Multiple dose pharmacokinetics profile for AZD8848 and its acid metabolite (AZ12432045) combined and, if possible, for AZD8848 alone in plasma | Plasma: From Days 1 and 22, pre-dose, 5, 10, 20, 30, 45, 60, 90 min, 2, 3, 4, 6, 8 and 24 hrs post dose
  PK parameters: AUC accumulation ratio and Cmax accumulation ratio
Pharmacodynamic effect after multiple doses of inhaled AZD8848 by assessment of the CXCL10 biomarker concentration in plasma | From Days 1 and 22, pre-dose, 24 and 48 hrs post dose. One sample 7 to 13 days post last dose.
  Pharmacodynamic effect: CXCL10 concentration and change-from-baseline ratios in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Tim Mant, BSc, MB BS, MRCP, FRCP, FFPM, Principal Investigator — Quintiles Drug Research Unit at Guy's Hospital, 6 Newcomen Street London SE1 1YR UK; Aray Aggarwal, Study Chair — AstraZeneca Pharmaceuticals 35 Gathouse Drive, Waltham, Ma 02451 United States
Locations (1):
- Research Site, London, United Kingdom

REFERENCES:
- [Derived] Delaney S, Biffen M, Maltby J, Bell J, Asimus S, Aggarwal A, Kraan M, Keeling D. Tolerability in man following inhalation dosing of the selective TLR7 agonist, AZD8848. BMJ Open Respir Res. 2016 Feb 23;3(1):e000113. doi: 10.1136/bmjresp-2015-000113. eCollection 2016. PMID 26933507
- See also: Study Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1661&filename=D0542C00002_Study_Synopsis.pdf